CLINICAL TRIAL: NCT06110702
Title: Randomized Trial on the Effects of an EMDR Intervention on Traumatic and Obsessive Symptoms During the COVID19 Quarantine: a Psychometric Study
Brief Title: Effects of an EMDR Intervention on Traumatic and Obsessive Symptoms
Acronym: MDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Andrea Poli, Research Fellow, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDL-01
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Adult ALL; Post-traumatic Stress Disorder; Obsessive-Compulsive Disorder; Disgust; Guilt; Shame
Keywords: PTSD; OCD; Disgust; Guilt; Shame; Body; EMDR
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-week EMDR Intervention (Experimental): Phase 1: The therapist and client develop a secure working relationship. The client's history is discussed and a treatment plan is developed.
  Phase 2: The therapist explains the EMDR therapy process. Phase 3: The target event is identified. Baseline measures are set using the Subjective Units of Disturbance (SUD) and the Validity of Cognition (VOC) scale.
  Phase 4: Desensitization, sounds, or taps are begun while focusing on the traumatic event until the client's SUD reduces to zero.
  Phase 5: The client associates and strengthens a positive belief with the target event until it feels true.
  Phase 6: The client is asked to hold in mind the target event and the positive belief while scanning the body.
  Phase 7: Reprocessing is complete when the client feels neutral about it (SUD=0, VOC=7), and the body is clear of disturbance.
  Phase 8: The client and therapist discuss processed memories to ensure that distress is low and that the positive cognition is strong.
  Interventions: Behavioral: EMDR
- Control condition - No intervention (No Intervention): The control group will follow routine daily activities

INTERVENTIONS:
Behavioral: EMDR — Eye movement Desensitization and Reprocessing (as described in the 8-phases protocol), administered both online or in presence.
  Arms: 8-week EMDR Intervention

SUMMARY:
The Eye Movement Desensitization and Reprocessing Protocol (EMDR) was first developed by Francine Shapiro in 1987 and can be adapted for online and in presence administration. The aim of this study is to assess if a EMDR program (administered both online and in presence, depending on different conditions of patients) may help people recruited from general population suffering from COVID19 second (November 2021 to February 2022) and third (March 2022 to May 2022) quarantine in improving post-traumatic stress (PTSD) and obsessive-compulsive-related (OCD) symptoms, as well as disgust, guilt, shame and their subjective unit of distress (SUD) and validity of cognition (VoC) levels.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 75 years
2. Participants experienced a full COVID19 pandemic-related quarantine during red zones of the second and third lockdowns in Italy
3. Participants have reasonable comprehension of spoken and written Italian language
4. Participants have an adequate understanding of Italian

Exclusion Criteria:

1. Concurrent enrollment in other intervention trials
2. Participants that already experienced EMDR therapy in the past

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Post-Traumatic Stress Symptoms - Pre-intervention | IES-R is measured immediately before the 8-week EMDR intervention
  Post-Traumatic symptoms are measured using the Impact of Event Scale-Revised (IES-R). The scale ranges from a minimum value of 0 to a maximum value of 88. Lower Likert score means a better outcome
Obsessive-Compulsive Symptoms - Pre-intervention | DOCS is measured immediately before the 8-week EMDR intervention
  Obsessive-Compulsive symptoms are measured using the Dimensional Obsessive-Compulsive Scale (DOCS). The scale ranges from a minimum value of 0 to a maximum value of 80. Lower Likert score means a better outcome
Body Perception - Pre-intervention | BPQ-22 is measured immediately before the 8-week EMDR intervention
  Body Perception is measured using the Body Perception Questionnaire-22 (BPQ-22). The scale ranges from a minimum value of 22 to a maximum value of 66. Lower Likert score means a better outcome
Guilt and Shame - Pre-intervention | GASP is measured immediately before the 8-week EMDR intervention
  Guilt and Shame are measured using the Guilt and Shame Proneness Scale (GASP). The scale ranges from a minimum value of 16 to a maximum value of 112. Lower Likert score means a better outcome
Disgust - Pre-intervention | TDDS is measured immediately before the 8-week EMDR intervention
  Disgust is measured using the Three Domain of Disgust Scale (TDDS). The scale ranges from a minimum value of 0 to a maximum value of 126. Lower Likert score means a better outcome
Mental Contamination - Pre-intervention | VOCI-MC is measured immediately before the 8-week EMDR intervention
  Mental Contamination is measured using the Vancouver Obsessional Compulsive Inventory-Mental Contamination scale (VOCI-MC). The scale ranges from a minimum value of 0 to a maximum value of 80. Lower Likert score means a better outcome
Post-Traumatic Stress Symptoms - Post-intervention | IES-R is measured immediately after the 8-week EMDR intervention
  Post-Traumatic symptoms are measured using the Impact of Event Scale-Revised (IES-R). The scale ranges from a minimum value of 0 to a maximum value of 88. Lower Likert score means a better outcome
Obsessive-Compulsive Symptoms - Post-intervention | DOCS is measured immediately after the 8-week EMDR intervention
  Obsessive-Compulsive symptoms are measured using the Dimensional Obsessive-Compulsive Scale (DOCS). The scale ranges from a minimum value of 0 to a maximum value of 80. Lower Likert score means a better outcome
Body Perception - Post-intervention | BPQ-22 is measured immediately after the 8-week EMDR intervention
  Body Perception is measured using the Body Perception Questionnaire-22 (BPQ-22). The scale ranges from a minimum value of 22 to a maximum value of 66. Lower Likert score means a better outcome
Guilt and Shame - Post-intervention | GASP is measured immediately after the 8-week EMDR intervention
  Guilt and Shame are measured using the Guilt and Shame Proneness Scale (GASP). The scale ranges from a minimum value of 16 to a maximum value of 112. Lower Likert score means a better outcome
Disgust - Post-intervention | TDDS is measured immediately after the 8-week EMDR intervention
  Disgust is measured using the Three Domain of Disgust Scale (TDDS). The scale ranges from a minimum value of 0 to a maximum value of 126. Lower Likert score means a better outcome
Mental Contamination - Post-intervention | VOCI-MC is measured immediately after the 8-week EMDR intervention
  Mental Contamination is measured using the Vancouver Obsessional Compulsive Inventory-Mental Contamination scale (VOCI-MC). The scale ranges from a minimum value of 0 to a maximum value of 80. Lower Likert score means a better outcome

SECONDARY OUTCOMES:
Anxiety Symptoms - Pre-intervention | DASS-21 is measured immediately before the 8-week EMDR intervention
  Anxiety symptoms are measured using the Depression Anxiety Stress Scales (DASS-21).The scale ranges from a minimum value of 0 to a maximum value of 63. Lower Likert score means a better outcome
Depression Symptoms - Pre-intervention | DASS-21 is measured immediately before the 8-week EMDR intervention
  Depression symptoms are measured using the Depression Anxiety Stress Scales (DASS-21). The scale ranges from a minimum value of 0 to a maximum value of 63. Lower Likert score means a better outcome
General distress symptoms - Pre-intervention | DASS-21 is measured immediately before the 8-week EMDR intervention
  General distress symptoms are measured using the Depression Anxiety Stress Scales (DASS-21). The scale ranges from a minimum value of 0 to a maximum value of 63. Lower Likert score means a better outcome
Anxiety Symptoms - Post-intervention | DASS-21 is measured immediately after the 8-week EMDR intervention
  Anxiety symptoms are measured using the Depression Anxiety Stress Scales (DASS-21). The scale ranges from a minimum value of 0 to a maximum value of 63. Lower Likert score means a better outcome
Depression Symptoms - Post-intervention | DASS-21 is measured immediately after the 8-week EMDR intervention
  Depression symptoms are measured using the Depression Anxiety Stress Scales (DASS-21). The scale ranges from a minimum value of 0 to a maximum value of 63. Lower Likert score means a better outcome
General distress symptoms - Post-intervention | DASS-21 is measured immediately after the 8-week EMDR intervention
  General distress symptoms are measured using the Depression Anxiety Stress Scales (DASS-21). The scale ranges from a minimum value of 0 to a maximum value of 63. Lower Likert score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Poli, PsyD, Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
Raw data are available on request.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Miccoli M, Poli A. Randomized trial on the effects of an EMDR intervention on traumatic and obsessive symptoms during the COVID-19 quarantine: a psychometric study. Front Psychiatry. 2024 Jun 26;15:1369216. doi: 10.3389/fpsyt.2024.1369216. eCollection 2024. PMID 38988736